CLINICAL TRIAL: NCT06822088
Title: Effects of Esketamine on Oxygenation and Quality of Recovery in Patients Undergoing Thoracoscopic Surgery
Acronym: OLV;Esk
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jinqiao Qian (Other)
Responsible Party: Sponsor-Investigator, Jinqiao Qian, Professor, First Affiliated Hospital of Kunming Medical University
Organization: First Affiliated Hospital of Kunming Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: (2024)ethical review L No.122; CXPJJH124001-19 (Other Grant/Funding Number: Hubei Chen xiaoping Science and Technology Development Foudation)
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Esketamine; One-lung Ventilation; Oxygenation Indices
Keywords: esketamine; one-lung ventilation; Oxygenation; Intrapulmonary shunt fraction; Lung protection
MeSH Terms: interventions — Esketamine; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Esketamine (Experimental): In Group E, 0.2mg/kg esketamine was infused intravenously before the induction of anesthesia for 10 min, and then maintained at 0.15 mg·kg-1·h-1 until 30 minutes before the end of the surgery.
  Interventions: Drug: Esketamine
- Dexmedetomidine (Active Comparator): Group D was given 1 ug/kg of dexmedetomidine 10min before surgery, and maintained at 0.4 ug/kg*h after intubation until 30min before the end of surgery
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator): Group C continued to pump the same amount of normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Esketamine — A total of 126 patients undergoing thoracoscopic surgery under elective general anesthesia were randomly divided into three groups: normal saline group (group C), dexmedetomidine group (group D), eschloroacetone group (group E) and dexmedetomidine group (group D), with 42 cases in each group. Group C was continuously injected with the same amount of normal saline, group D was given dextrometin 1 ug/kg load 10min before surgery, and maintained at 0.4 ug/kg*h after intubation until 30min before the end of surgery. Group E was given esketamine 0.2 mg/kg 10min before surgery, and maintained at 0.15 mg/kg*h after intubation until 30min before surgery. Other anesthetic induction and maintenance drugs were consistent among the three groups.
  Arms: Esketamine
Drug: Dexmedetomidine — group D was given Dexmedetomidine 1 ug/kg load 10min before surgery, and maintained at 0.4 ug/kg*h after intubation until 30min before the end of surgery.
  Arms: Dexmedetomidine
Drug: Normal Saline — Group C was continuously injected with the same amount of normal saline,
  Arms: Normal saline

SUMMARY:
A total of 126 patients undergoing elective thoracoscopic surgery under general anesthesia were randomly divided into three groups: normal saline group (Group C), dexmedetomidine group (Group D), and esketamine group (Group E),with 42 patients in each group.In Group C,an equal volume of normal saline was continuously infused. In Group D,a loading dose of dexmedetomidine (1 μg/kg) was administered 10 min before induction of anesthesia, followed by a continuous infusion at a rate of 0.4 μg·kg-1·h-1 until 30 minutes before the end of the surgery. In Group E, 0.2mg/kg esketamine was infused intravenously before the induction of anesthesia for 10 min, and then maintained at 0.15 mg·kg-1·h-1 until 30 minutes before the end of the surgery. The primary outcome measures of this study were the oxygenation index (OI) at the following time points: before one-lung ventilation (OLV) (T1), 30 minutes after OLV initiation (T2), and 60 minutes after OLV initiation (T3). The secondary outcome measures included: (1)The duration of OLV, blood loss, fluid infusion volume, the dosages of propofol, remifentanil and vasoactive drugs(ephedrine and atropine) were recorded in each group.(2)Heart rate (HR) and mean arterial pressure (MAP) were recorded at the following time points: upon entering the operating room (T0), before OLV (T1), 30 minutes after OLV initiation (T2), 60 minutes after OLV initiation (T3), before extubation (T4), and 5 minutes after extubation (T5).(3)Blood gas anlaysis parameters,airway plateau pressure,tidal volume and positive end-expiratory pressure were recorded from T1 to T3，and dynamic lung compliance and intrapulmonary shunt fraction were calculated.(4) White blood cell counts, neutrophil percentage,and C-reactive protein (CRP) levels were recorded preoperatively and 24 hours postoperatively.(5)Postoperative pain was evaluated using the visual analogue score (VAS) at 2, 6, 12, and 24 hours after surgery, and the number of patients requiring rescue analgesia in each group was recorded. The occurrence of postoperative adverse reactions and postoperative pulmonary complications (PCCs) within one week after surgery were recorded. The postoperative quality of recovery was evaluated using the QOR-15 scale at 24 and 48 hours after surgery,and the postoperative hospital stay was recorded.

DETAILED DESCRIPTION:
Objective：To investigate the effects of esketamine on oxygenation during one-lung ventilation (OLV) and the quality of recovery in patients undergoing thoracoscopic surgery . This study aims to systematically evaluate the clinical efficacy of esketamine and explore its potential advantages in thoracoscopic procedures. The findings are expected to provide new insights into optimizing lung protection strategies during OLV, thereby enhancing perioperative management and improving outcomes for patients undergoing thoracoscopic surgery.

Method：A total of 126 patients undergoing elective thoracoscopic surgery under general anesthesia were randomly divided into three groups: normal saline group (Group C), dexmedetomidine group (Group D), and esketamine group (Group E),with 42 patients in each group.In Group C,an equal volume of normal saline was continuously infused. In Group D,a loading dose of dexmedetomidine (1 μg/kg) was administered 10 min before induction of anesthesia, followed by a continuous infusion at a rate of 0.4 μg·kg-1·h-1 until 30 minutes before the end of the surgery. In Group E, 0.2mg/kg esketamine was infused intravenously before the induction of anesthesia for 10 min, and then maintained at 0.15 mg·kg-1·h-1 until 30 minutes before the end of the surgery. The primary outcome measures of this study were the oxygenation index (OI) at the following time points: before one-lung ventilation (OLV) (T1), 30 minutes after OLV initiation (T2), and 60 minutes after OLV initiation (T3). The secondary outcome measures included: (1)The duration of OLV, blood loss, fluid infusion volume, the dosages of propofol, remifentanil and vasoactive drugs(ephedrine and atropine) were recorded in each group.(2)Heart rate (HR) and mean arterial pressure (MAP) were recorded at the following time points: upon entering the operating room (T0), before OLV (T1), 30 minutes after OLV initiation (T2), 60 minutes after OLV initiation (T3), before extubation (T4), and 5 minutes after extubation (T5).(3)Blood gas anlaysis parameters,airway plateau pressure,tidal volume and positive end-expiratory pressure were recorded from T1 to T3，and dynamic lung compliance and intrapulmonary shunt fraction were calculated.(4) White blood cell counts, neutrophil percentage,and C-reactive protein (CRP) levels were recorded preoperatively and 24 hours postoperatively.(5)Postoperative pain was evaluated using the visual analogue score (VAS) at 2, 6, 12, and 24 hours after surgery, and the number of patients requiring rescue analgesia in each group was recorded. The occurrence of postoperative adverse reactions and postoperative pulmonary complications (PCCs) within one week after surgery were recorded. The postoperative quality of recovery was evaluated using the QOR-15 scale at 24 and 48 hours after surgery,and the postoperative hospital stay was recorded.

Background：According to the cancer statistics report released by the American Cancer Society in 2024, about one in five people will develop cancer in lifetime, and about one in nine men and one in twelve women will die of cancer. Lung cancer is the most commonly occurring cancer worldwide (accounting for 1.4% of all new cases) and is also the leading cause of cancer death (accounting for 18.7% of total cancer deaths), nearly twice second leading cause of cancer death.At present, surgery is the preferred treatment for early-stage lung cancer, and timely and effective surgical treatment can effectively reduce risk of tumor recurrence and metastasis, and improve the survival rate of patients.With the continuous development of modern medical technology, the surgical approach for lung cancer has evolved from traditional open thoracotomy to video-assisted thor surgery (VATS). As a minimally invasive surgery, VATS has many advantages, such as small incision, rapid postoperative recovery, and fewer postoperative. VATS usually requires the use of a double-lumen endobronchial tube (DLT) or a bronchial blocker to perform one-lung (OLV) on the nonoperative side. OLV is a ventilation technique that separates the ventilation pathways of both sides at the level of the carina. The is to collapse the surgical side of the lung and protect the nonoperative side of the lung from contamination, while also facilitating the exposure of the surgical field and reducing the of surgical complications.However,during OLV, the atelectatic lung, although not ventilated, still has blood flow through it, and this blood is not oxygenated, in a mismatch in the ventilation/perfusion ratio (VA/Q), leading to an increase in intrapulmonary shunting and a decrease in oxygenation, which in leads to hypoxemia.Secondly, thoracic surgery is generally performed in the lateral position, and due to the influence of gravity, the patient's ventilation and blood flow distribution uneven, with the shunt fraction reaching as high as 40-50%.Hypoxia and ischemic injury as well as cellular damage can be caused by insufficient ventilation. During the process of restoring blood supply, will also aggravate cellular damage, cause pathological and physiological changes in the lung, trigger ischemia-reperfusion injury, hypoxemia, and then acute inflammatory response oxidative stress response, causing acute injury to a variety of organs. In recent years, with the implementation of lung-protective ventilation strategy, the application and popularization fiberoptic bronchoscopy and video double-lumen bronchial intubation, the incidence of hypoxemia has decreased, but the incidence in thoracic is still 10% to 25%.Strategies to improve hypoxemia include pharmacological reduction of intrapulmonary shunt, improvement of ventilation-perfusion mismatch, and improvement of strategies . The strategy of ventilating the surgical lung is not conducive to the collapse of the surgical lung during thoracoscopy, affecting the exposure of the field. At present, the use of pharmacological intervention is a new idea in the study of improving hypoxemia during OLV of thoracoscopy.

Esketamine, as a new type of intravenous anesthetic, is a high-affinity N-methyl-D-aspartate (NA) receptor non-competitive inhibitor. As the S-enantiomer of ketamine, it has a similar mechanism of action to ketamine, but with a higher for the NMDA receptor and a potency twice that of ketamine. Therefore, compared with traditional ketamine, a smaller dose can achieve the desired anesthetic effect while reducing the incidence of psychotropic side effects. Its effects can produce analgesia, sedation, anti-inflammation, anti-depression, mild respiratory depression and mild circulatory excitation.Esketamine can directly act on the airway smooth muscle, dilate the bronchi and relax the airway through voltage-dependent L-type calcium, effectively relieve bronchospasm, reduce airway resistance, improve lung compliance, and improve ventilation and gas exchange function.Meanwhile, esketamine can inhibit the release of inflammatory cells stimulated by oxygen free radicals, reduce the secretion of various cytokines such as TNFα, IL-6 and IL-8 by white blood cells, inhibit the expression of adhesion factors on the surface of neutrophils and the activity of induc nitric oxide synthase, and promote the secretion of anti-inflammatory cytokines, which can play a multi-level antagonistic role in inflammation.Many studies have suggested that esmolol may be a potential drug intervention to improve perioperative oxygenation.

Dexmedetomidine is a highly selective α2-adrenergic receptor agonist, which mainly produces sedative, analgesic,-anxiety, and sympatholytic effects by acting on the central nervous system, peripheral nervous system, and other organ tissues.Recent studies have shown that dexmedetomidine can reduce the inflammatory response and oxidative stress of thoracic surgery by reducing the levels of plasma,-6, IL-8, TNF-α, and lipid peroxidation in patients, improve the expression of aquaporin in lung tissue of thoracic, increase the concentration of nitric oxide in the blood, dilate the pulmonary vessels on the ventilated side, and effectively reduce intrapulmonary shunting and oxygenation.In addition, dexmedetomidine can directly enhance HPV by targeting α2B receptors in vascular smooth muscle and inducing vasoconstriction in the nonventilated lung, improving the intraoperative oxygenation index, reducing dead space ventilation, improving the dynamic compliance of the lung, and reducing the incidence of postoperative, playing an important role in lung protection.

Based on the above research on esmolol, this study will explore the effects of esmolol on patients' oxygenation and intrapul shunting during single-lung ventilation in thoracoscopy surgery on the basis of previous research, and further clarify the advantages of esmolol in thoracoscopy surgery and provide new clinical basis for optimizing the lung protection strategy during single-lung ventilation in thoracoscopy surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracoscopic surgery under elective general anesthesia in the First Affiliated Hospital of Kunming Medical University;
* Age 18-65 years old;
* BMI18~30 kg/m2;
* American Society of Anesthesiologistsgrade I~III;
* No contraindications to drugs;
* All patients and their families agreed to participate in this study and signed informed consent

Exclusion Criteria:

* Patients with severe sinus bradycardia (heart rate <50 beats/min) and atrioventricular block;
* Respiratory infection and non-steroidal anti-inflammatory drugs or hormone drugs taken within 2 weeks before surgery;
* severe liver and kidney dysfunction and immune system diseases, uncontrolled hypertension, diabetes;
* History of preoperative chemoradiotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Index；Quality of postoperative recovery | 7 days
  Esketamine can improve oxygenation during one-lung ventilation in patients undergoing thoracoscopy, producing a lung-protective effect; at the same, it improves the quality of postoperative recovery in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2025.03.01-2026.03.01

REFERENCES:
- [Background] Shi J, Yu T, Song K, Du S, He S, Hu X, Li X, Li H, Dong S, Zhang Y, Xie Z, Li C, Yu J. Dexmedetomidine ameliorates endotoxin-induced acute lung injury in vivo and in vitro by preserving mitochondrial dynamic equilibrium through the HIF-1a/HO-1 signaling pathway. Redox Biol. 2021 May;41:101954. doi: 10.1016/j.redox.2021.101954. Epub 2021 Mar 21. PMID 33774474
- [Background] Xie Y, Jiang W, Zhao L, Wu Y, Xie H. Effect of dexmedetomidine on perioperative inflammation and lung protection in elderly patients undergoing radical resection of lung cancer. Int J Clin Exp Pathol. 2020 Oct 1;13(10):2544-2553. eCollection 2020. PMID 33165407
- [Background] Cai SY, Liu A, Xie WX, Zhang XQ, Su B, Mao Y, Weng DG, Chen ZY. Esketamine mitigates mechanical ventilation-induced lung injury in chronic obstructive pulmonary disease rats via inhibition of the MAPK/NF-kappaB signaling pathway and reduction of oxidative stress. Int Immunopharmacol. 2024 Sep 30;139:112725. doi: 10.1016/j.intimp.2024.112725. Epub 2024 Jul 25. PMID 39059100
- [Background] Tu W, Yuan H, Zhang S, Lu F, Yin L, Chen C, Li J. Influence of anesthetic induction of propofol combined with esketamine on perioperative stress and inflammatory responses and postoperative cognition of elderly surgical patients. Am J Transl Res. 2021 Mar 15;13(3):1701-1709. eCollection 2021. PMID 33841692
- [Background] Campos JH, Feider A. Hypoxia During One-Lung Ventilation-A Review and Update. J Cardiothorac Vasc Anesth. 2018 Oct;32(5):2330-2338. doi: 10.1053/j.jvca.2017.12.026. Epub 2017 Dec 19. No abstract available. PMID 29361458
- [Background] Durkin C, Romano K, Egan S, Lohser J. Hypoxemia During One-Lung Ventilation: Does It Really Matter? Curr Anesthesiol Rep. 2021;11(4):414-420. doi: 10.1007/s40140-021-00470-5. Epub 2021 Jul 7. PMID 34254003
- [Background] Lumb AB, Slinger P. Hypoxic pulmonary vasoconstriction: physiology and anesthetic implications. Anesthesiology. 2015 Apr;122(4):932-46. doi: 10.1097/ALN.0000000000000569. PMID 25587641
- [Background] Archer SL, Dunham-Snary KJ, Bentley R, Alizadeh E, Weir EK. Hypoxic Pulmonary Vasoconstriction: An Important Component of the Homeostatic Oxygen Sensing System. Physiol Res. 2024 Nov 29;73(S2):S493-S510. doi: 10.33549/physiolres.935431. PMID 39589299
- [Background] Alday E, Nieves JM, Planas A. Oxygen Reserve Index Predicts Hypoxemia During One-Lung Ventilation: An Observational Diagnostic Study. J Cardiothorac Vasc Anesth. 2020 Feb;34(2):417-422. doi: 10.1053/j.jvca.2019.06.035. Epub 2019 Jun 28. PMID 31362907
- [Background] Nierengarten MB. Global cancer statistics 2022: The report offers a view on disparities in the incidence and mortality of cancer by sex and region worldwide and on the areas needing attention. Cancer. 2024 Aug 1;130(15):2568. doi: 10.1002/cncr.35444. No abstract available. PMID 39032060